CLINICAL TRIAL: NCT02652143
Title: Does in Vivo Culture of Pre-cleavage Stage Embryo Reduce the Incidence of Aneuploidy? A Sibling Oocyte, Prospective, Multi-centric, Randomized, Open Study, Clinical Study in Subjects With Subfertility Undergoing Assisted Reproductive Medical Treatment
Brief Title: Does in Vivo Culture of Pre-cleavage Stage Embryo Reduce the Incidence of Aneuploidy?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to difficult recruitment
Sponsor: Anecova SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCVd20H
Record Dates: First submitted 2016-01-07; First posted 2016-01-11 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Infertility; Reproductive Sterility
Keywords: in vivo culture
MeSH Terms: conditions — Infertility | interventions — Equipment and Supplies; In Vitro Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sibling oocytes in vivo (Experimental): randomized oocytes assigned to in vivo culture
  Interventions: Device: AneVivo (Medical device for in vivo culture of embryos)
- sibling oocyte in vitro (Active Comparator): randomized oocytes assigned to in vitro culture
  Interventions: Other: comparator for embryo culture in vitro

INTERVENTIONS:
Device: AneVivo (Medical device for in vivo culture of embryos)
  Other Names: Anecova
  Arms: sibling oocytes in vivo
Other: comparator for embryo culture in vitro
  Arms: sibling oocyte in vitro

SUMMARY:
This Clinical Study has been designed to assess and compare the impact of in vitro or in vivo culture conditions on the euploidy of sibling blastocysts.

DETAILED DESCRIPTION:
As soon as the very first minute of the fertilization process, very important biological events, critical for the future developmental competency of the embryo are taking place.

These biological events, after the sperm cell entry in the oocyte cytoplasm and prior to the first cleavage, include: the completion of the meiosis, the exclusion of the second polar body, the pronuclei formation, the replication of the male and female DNA and the chromosome segregation on the newly formed mitotic spindle.

If any of these events is aberrant, one or both of the two daughter cells and their descendants may carry chromosomal anomalies. In other words an uneven first cleavage in size or in content is associated with chromosomal abnormality and aneuploidy.

In vivo all these events occur in a natural environment where the presence of specific molecules and of a dynamic and physiological environment might be an advantage over in vitro culture conditions to ensure optimal cellular functions.

Preliminary data from the pilot study have shown a higher proportion of euploid embryos for sibling oocytes cultured in vivo vs. in vitro. Moreover, in animal models, in vivo cultured embryos have been described with significant reduction of aneuploidies and with differences in the gene expression levels patterns when compared to in vitro cultured embryos. There is also growing evidence that the culture conditions of human pre-implantation embryos can affect the gene expression regulation with measurable effects on embryos and on newborn children.

The investigators hypothesis is that in vivo produced embryos might have a higher percentage of euploidy when compared to their siblings cultured in vitro.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent by the subject and her partner
* Women, aged between 18 and 38 years (up to 38th birthday)
* ≤ 2 previous stimulation cycles
* Routinely measured hormonal levels within normal range (i.e. FSH, LH, E2, PRL)
* No uterine or ovarian anatomical abnormalities and/or alterations that would compromise device delivery or function in the uterus as demonstrated by ultrasound and trial insertion
* 19 ≤ BMI ≤ 29 kg/m2

Exclusion Criteria:

* History of previous moderate or severe ovarian hyperstimulation syndrome (OHSS)
* Severe endometriosis
* Any active infection that would contraindicate ART, at the discretion of the investigator
* Severe male factor in the partner (cryptozoospermia or non-obstructive azoospermia)

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Euploidy status after a biopsy on all viable day 5 embryos | 1 week
  full genome analysis on 24 chromosomes

SECONDARY OUTCOMES:
Implantation rate | 9 weeks
  number of gestational sac per transferred embryos
Pregnancy rate | 9 weeks
  beating heart

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Ferrando, MD, Principal Investigator — IVI Bilbao
Locations (1):
- Ivi Bilbao, Bilbao, Spain

IPD SHARING:
Plan to Share IPD: Undecided